CLINICAL TRIAL: NCT00001788
Title: Molecular Basis of Primary Immunodeficiencies
Brief Title: Genetic Basis of Primary Immunodeficiencies
Status: Terminated | Type: Observational
Why Stopped: Investigator left NIH
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990004; 99-AR-0004
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Immunologic Deficiency Syndrome
Keywords: Cytokine; Stat; Jak; IL-12; Mutation; Immunodeficiency
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Samples with and without DNA are being retained. These include patient white cells, patient dermal fibroblasts, patient iPS cells and patient serum.

GROUPS / COHORTS (1):
- 1: patients with primary immunodeficiency disorders

SUMMARY:
The purpose of this study is to evaluate patients with primary immunodeficiency disorders to identify patients with mutations of the genes for the following proteins: Jak3, STAT1, STAT4, interleukin-7, interleukin-7 receptor, interleukin-12 receptor subunits, and others.

Patients will undergo screening history, physical examination, and clinical laboratory evaluation at referring institutions and tissue samples, or cell lines will be sent to the NIH. We will establish cell lines if necessary, prepare DNA and RNA for molecular genetic analysis and study cytokine signal transduction in patient cell lines.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate patients with primary immunodeficiency disorders to identify patients with mutations of the genes for the following proteins: Jak3, STAT1, STAT4, interleukin-7, interleukin-7 receptor, interleukin-12 receptor subunits, and others. Patients will undergo screening history, physical examination, and clinical laboratory evaluation at referring institutions and tissue samples, or cell lines will be sent to the NIH. We will establish cell lines if necessary, prepare DNA and RNA for molecular genetic analysis and study cytokine signal transduction in patient cell lines.

ELIGIBILITY:
* INCLUSION CRITERIA:

Samples from patients with known or suspected primary immunodeficiencies, including those treated with stem cell transplants or gene correction therapy, and their families will be accepted worldwide primarily from tertiary care centers that treat patients with such immunodeficiencies.

Such patients will have documented evidence of either opportunistic infection, recurrent infection, or unusually severe responses to infectious agents that cause mild illness in unaffected individuals. In selected cases, at the discretion of the investigators, samples for testing will be obtained from consenting adult relatives of affected individuals.

Either patient-derived B cell lines or primary blood samples will be accepted although in some cases buccal swabs will also be accepted.

Blood samples may be obtained from unaffected children.

Additionally; patients with particularly interesting clinical presentations (e.g. adults with possible attenuated immunodeficiency) may be seen for outpatient visits at the NIH Clinical Center for evaluation.

Infants with SCID or other primary immunodeficiency will not be seen; their physicians will care them for and only clinical material will be sent on such patients.

Medically stable patients with mild to moderate immunodeficiency may be seen at the NIH.

We will encourage the participation of women and members of minority groups in this study.

EXCLUSION CRITERIA:

Inability to provide informed consent.

A presence of any medical condition that would, in the opinion of the investigators, confuse the interpretation of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: (1) Patients will be examined at the NIH where relevant samples will be collected for analysis.(2) Patients will be examined by outside physicians and relevant patient history and physical results and samples sent to the NIH for evaluation.(3) Patients samples may be sent to us from Duke University Medical Center, a tertiary center with extensive experience in diagnosis and treatment of primary immunodeficiencies.(4) In the future, patient samples may be sent from other tertiary care centers not identified at this time.(5) Family members of patients with primary immunodeficiencies, if they or their parents/guardians request, may be evaluated at the discretion of the investigators.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2011-08-21 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Natural History of Immunologic Deficiency Syndrome | Enrollment with follow-up
  The objectives of the study are: (1) To identify new patients with Jak3 deficiency to determine the range of mutations that occur, to study these mutations in in vitro assays and to relate these findings to the clinical presentation. We will also try to develop improved assays for the diagnosis of Jak3 deficiency. (2) To analyze the function of lymphoid and myeloid cells from patients who have undergone stem cell transplants for Jak3- and XSCID (3) To analyze patients with TB+SCID without mutations of Jak3 and c for mutations in IL- 7, IL-7 receptor genes. (4) To analyze patients with defects in cell-mediated immunity to try to identify patients with mutations of the genes encoding IL-12 subunits, IL-12 receptor subunits and the transcription factors Stat1, Stat 4 and IRF.
Natural History of Immunologic Deficiency Syndrome | Enrollment with follow-up
  The objectives of the study are: (5) To analyze patients, including their tissues and cells, with defects in innate immunity, adaptive immunity, or both who clinically present with features suggestive of NEMO Syndrome or NEMO-like syndrome to identify individuals with mutations in IKK (NEMO), IB, and other genes that modify the expression and function of NFB family members.
Natural History of Immunologic Deficiency Syndrome | Enrollment with follow-up
  The objectives of the study are: (6) To perform whole genome, exome, or chemical analysis of genes in selected patients and family members to discover new primary immunodeficiency related genes. Whole genome, exome, or other gene analysis will be done to determine which particular genetic variations can cause the various primary immunodeficiencies such as JAK3 deficiency or NEMO Syndrome. We also seek to study whether particular variations are associated with more or less severe illness, or with specific types of symptoms, to understand the basic mechanism by which these altered genes cause cells to function differently, and to identify other genes causing SCID or NEMO-like syndrome. In order to do this, we need blood specimens (or cells from inside the cheek) from patients and their families. We will use these samples to identify which, if any, abnormality is present in the patient s genes, and to study the behavior of immune cells in vitro.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Colbert, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Lee Y, Wessel AW, Xu J, Reinke JG, Lee E, Kim SM, Hsu AP, Zilberman-Rudenko J, Cao S, Enos C, Brooks SR, Deng Z, Lin B, de Jesus AA, Hupalo DN, Piotto DG, Terreri MT, Dimitriades VR, Dalgard CL, Holland SM, Goldbach-Mansky R, Siegel RM, Hanson EP. Genetically programmed alternative splicing of NEMO mediates an autoinflammatory disease phenotype. J Clin Invest. 2022 Mar 15;132(6):e128808. doi: 10.1172/JCI128808. PMID 35289316
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1999-AR-0004.html